CLINICAL TRIAL: NCT05187559
Title: Effectiveness of a Neuromuscular Exercise Program and Visual Feedback in the Management of Body Position During Standing and Walking for Patients With Stroke During the Second Stage of Rehabilitation
Brief Title: Effectiveness of a Neuromuscular Exercise Program and Visual Feedback in the Management of Body Position for Stroke Survivors
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Lithuanian University of Health Sciences (Other)
Responsible Party: Principal Investigator, Toma Steponkienė, PhD student, Lecturer, Lithuanian University of Health Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RK-NRB-TS-01
Record Dates: First submitted 2021-11-22; First posted 2022-01-12 (Actual); Last update posted 2022-01-12 (Actual); Status verified 2022-01

CONDITIONS: Brain Ischemia; Stroke, Ischemic
Keywords: Brain Ischemia; Stroke; Balance; Gait; Physiotherapy; Physical Therapy; Visual Feedback
MeSH Terms: conditions — Brain Ischemia; Ischemic Stroke; Stroke

STUDY DESIGN:
Intervention Model Description: Two study groups, 60 patients per group. Patients will be randomly assigned to first of second study group.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- First Group (Experimental): Neuromuscular exercise program with standard physiotherapy with no visual feedback.
  Interventions: Other: Standard physiotherapy
- Second Group (Experimental): Neuromuscular exercise program with physiotherapy with visual feedback using Biodex platform
  Interventions: Device: Biodex Balance SD and Biodex Gait Trainer

INTERVENTIONS:
Other: Standard physiotherapy — Neuromuscular exercise program with standard physiotherapy with no visual feedback
  Arms: First Group
Device: Biodex Balance SD and Biodex Gait Trainer — Neuromuscular exercise program with physiotherapy with visual feedback using Biodex platform
  Arms: Second Group

SUMMARY:
The aim of the biomedical research is to evaluate the changes of body position management during standing and walking for stroke patients, using innovative training methods during the rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* Experienced an ischemic stroke for the first time;
* Middle-aged (44-59) and elderly (60-74) by WHO classification;
* Muscle strength of the lower extremities according to the Oxford scale is 3-5 points;
* Do not have any neglect;
* Mini Mental State Examination >12 points.

Exclusion Criteria:

* Experienced an ischemic stroke not for the first time;
* Had hip or knee replacement surgery's, which may affect gait;
* Muscle strength of the lower extremities according to the Oxford scale is 0-2 points;
* Have neglect;
* Mini Mental State Examination <12 points.

Ages: 44 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2021-12-01 (Actual); Primary Completion 2024-08-31 (Estimated); Study Completion 2024-08-31 (Estimated)

PRIMARY OUTCOMES:
Muscle strength by Oxford scale | Baseline
  Testing key muscles from the lower and upper extremities against the examiner's resistance and grading the patient's strength on a 0 (No contraction) to 5 (Movement against gravity with full resistance) scale.
Gait and Balance testing by Berg Scale | Baseline
  The Berg balance scale is used to objectively determine a patient's ability (or inability) to safely balance during a series of predetermined tasks. It consists of 14 items scored on an ordinal scale of 0 to 4 for a total of 56 points (a higher score indicates lower fall risk).
Timed Stand Up and Go Test | Baseline
  subjects are asked to rise from a standard armchair, walk to a marker 3 m away, turn, walk back, and sit down again. 314. The test is a reliable and valid test for quantifying functional mobility that may also be useful in following clinical change over time.
Recovery Locus of Control Scale | Baseline
  This scale contains 9 statements that are designed to evaluate the internal and external beliefs regarding the traumatic events that the patient has experienced.

SECONDARY OUTCOMES:
Limits of Stability Testing with Biodex SD (score) | Baseline - before enrolling 4 week training program and after 4 week training
  During test, patients must shift their weight to move the cursor from the center target to a colored target and back as quickly and with as little deviation as possible. Platform Setting- static. Direction control - overall. Faster and accurately- better.
Risk of Fall Testing with Biodex SD (score) | Baseline - before enrolling 4 week training program and after the whole training
  Test results are compared to age dependent normative data. Platform Setting - static. Test Trial Time 30 seconds in four positions: eyes opened narrow stance, eyes closed narrow stance, eyes opened closed feet stance, eyes closed stance. Patient's aged 54-71 years' normative scores are 0.9-3.7 scores, 72-89 years' normative scores are 2-4 scores, 36-53 years' normative scores are 0.7-3.1 scores, 17-35 years' normative scores are 0.7-2.1 scores. Change from baseline indicates a fall risk by scores.
Stance analysis with zebris FDM (score) | Baseline - before enrolling 4 week training program and after 4 week training
  Stance phase analysis (stance parameters and forces) - average load distribution under the feet is displayed in color. The color scale enables the load distribution to be quantified. The central point's show the centers of pressure (COP) over the time. The left and right points are the respective centers of pressure of the left and right contact areas. The area of the displayed confidence ellipse contains 95% of the COP's measuring points.
Gait analysis with zebris FDM (score) | Baseline - before enrolling 4 week training program and after 4 week training
  Analysis of gait geometry: Foot rotation(degree)
Gait analysis with zebris FDM (score) | Baseline - before enrolling 4 week training program and after 4 week training
  Analysis of gait geometry: Step length(cm)
Gait analysis with zebris FDM (score) | Baseline - before enrolling 4 week training program and after 4 week training
  Analysis of gait geometry:Stride length(cm)
Gait analysis with zebris FDM (score) | Baseline - before enrolling 4 week training program and after 4 week training
  Analysis of gait geometry: Step width(cm)
Gait analysis with zebris FDM (score) | Baseline - before enrolling 4 week training program and after 4 week training
  Analysis of gait phases: Stance phase(%)
Gait analysis with zebris FDM (score) | Baseline - before enrolling 4 week training program and after 4 week training
  Analysis of gait phases: Load response(%)
Gait analysis with zebris FDM (score) | Baseline - before enrolling 4 week training program and after 4 week training
  Analysis of gait phases: Single limb support(%)
Gait analysis with zebris FDM (score) | Baseline - before enrolling 4 week training program and after 4 week training
  Analysis of gait phases: Pre-Swing(%)
Gait analysis with zebris FDM (score) | Baseline - before enrolling 4 week training program and after 4 week training
  Analysis of gait phases: Swing phase(%)
Gait analysis with zebris FDM (score) | Baseline - before enrolling 4 week training program and after 4 week training
  Analysis of gait phases: Double stance phase(%)
Gait analysis with zebris FDM (score) | Baseline - before enrolling 4 week training program and after 4 week training
  Analysis of gait timing: Step time(sec)
Gait analysis with zebris FDM (score) | Baseline - before enrolling 4 week training program and after 4 week training
  Analysis of gait timing: Stride time(sec)
Gait analysis with zebris FDM (score) | Baseline - before enrolling 4 week training program and after 4 week training
  Analysis of gait timing: Cadence(steps/min)
Gait analysis with zebris FDM (score) | Baseline - before enrolling 4 week training program and after 4 week training
  Analysis of gait timing: Velocity(km/h)
Center of Pressure analysis during step cycles with zebris FDM (score) | Baseline - before enrolling 4 week training program and after 4 week training
  COP analysis (Butterfly parameters): Length of gait line(mm)
Center of Pressure analysis during step cycles with zebris FDM (score) | Baseline - before enrolling 4 week training program and after 4 week training
  COP analysis (Butterfly parameters): Single limb support line(mm)
Center of Pressure analysis during step cycles with zebris FDM (score) | Baseline - before enrolling 4 week training program and after 4 week training
  COP analysis (Butterfly parameters): Anterior/posterior position(mm)
Center of Pressure analysis during step cycles with zebris FDM (score) | Baseline - before enrolling 4 week training program and after 4 week training
  COP analysis (Butterfly parameters): Lateral symmetry(mm)
Center of Pressure analysis during step cycles with zebris FDM (score) | Baseline - before enrolling 4 week training program and after 4 week training
  COP analysis (Butterfly parameters): Max gait line velocity(cm/sec)
Center of Pressure analysis during step cycles with zebris FDM (score) | Baseline - before enrolling 4 week training program and after 4 week training
  COP analysis (Load change parameters): Time change heel to forefoot(sec)
Center of Pressure analysis during step cycles with zebris FDM (score) | Baseline - before enrolling 4 week training program and after 4 week training
  COP analysis (Load change parameters): Time change heel to forefoot(%)
Center of Pressure analysis during step cycles with zebris FDM (score) | Baseline - before enrolling 4 week training program and after 4 week training
  COP analysis (Load change parameters): Maximum force (Forefoot, Midfoot, Heel) (N)
Center of Pressure analysis during step cycles with zebris FDM (score) | Baseline - before enrolling 4 week training program and after 4 week training
  COP analysis (Load change parameters): Maximum pressure (Forefoot, Midfoot, Heel) (N/cm²)
Center of Pressure analysis during step cycles with zebris FDM (score) | Baseline - before enrolling 4 week training program and after 4 week training
  COP analysis (Load change parameters): Time maximum force (Forefoot, Midfoot, Heel)(% of stance)

CONTACTS AND LOCATIONS:
Overall Officials: Eglė Lendraitienė, PhD, Principal Investigator — Lithuanian University of Health Sciences
Locations (1):
- Toma Steponkienė, Kaunas, Lithuania

IPD SHARING:
Plan to Share IPD: No